CLINICAL TRIAL: NCT04497532
Title: The Influence of a Diet Suited for Gestational Diabetes on Amniotic Fluid Index in Patients Diagnosed With Idiopathic Polyhydramnios - a Randomized Controlled Trial
Brief Title: Influence of Diet on Pregnancy With Polyhydramnios
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Liliya Tamayev, Principal Investigator, Wolfson Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0152-19-WOMC
Record Dates: First submitted 2020-07-29; First posted 2020-08-04 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Polyhydramnios
MeSH Terms: conditions — Polyhydramnios | interventions — Diet

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Diet (Experimental)
  Interventions: Other: Diet as suited for gestational diabetes mellitus

INTERVENTIONS:
Other: Diet as suited for gestational diabetes mellitus — Diet that consists of complex carbohydrates, and a regimen that includes 6 meals per day, as tailored gor gestational diabetes.
  Arms: Diet

SUMMARY:
To evaluate the effect of a diet that is suited for gestational diabetes mellitus on amniotic fluid index in women with idiopathic polyhydramnios.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between 24-37 pregnancy weeks, singleton pregnancy, diagnosed with AFI at 95% or more by gestational age
* Express their consent to participate in the study and try to make the recommended dietary change for at least two consecutive weeks from the moment the guidelines are given.
* Without a medical indication for an immediate delivery

Exclusion Criteria:

* Medical recommendation for delivery within two weeks of diagnosis
* Condition of non-idiopathic amniotic fluid: gestational or pre-gestational diabetes, fetal malformation, proof of fetal infection
* Premature rupture or membranes
* Twins pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-03-20 (Estimated); Primary Completion 2022-12-20 (Estimated); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
Amniotic fluid index (AFI) after 2 weeks | Assess AFI two weeks after diet initiation
  AFI as measured in ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Liliya Tamayev, MD, Principal Investigator — Wolfson Medical Center

IPD SHARING:
Plan to Share IPD: No